CLINICAL TRIAL: NCT00423020
Title: Erythropoietin Prevention Trial of Coronary Restenosis and Cardiac Remodeling After Acute Myocardial Infarction (EPOC-AMI)
Brief Title: Anti-Restenosis After AMI by Erythropoietin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyoto Prefectural University of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPOC-AMI 2006
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2007-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Restenosis; erythropoietin; EPOC-AMI
MeSH Terms: interventions — Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin

SUMMARY:
The EPOC-AMI study is to assess the safety and the efficacy of systemic administration of erythropoietin for inhibition of neointimal hyperplasia after stent implantation in the patients with acute myocardial infarction

DETAILED DESCRIPTION:
Stents coated with sirolimus or paclitaxel have been shown to significantly reduce restenosis in selected coronary lesions. However, the potential risk of late stent thrombosis forces prolonged treatment of dual anti-platelet regimen to all the patients after implantation of drug eluting stents. Patients with acute myocardial infarction may have uncertain clinical characteristics, such as occult bleeding focus or further need for surgical procedures. Thus, bare metal stent is considerably alternative for primary PCI after AMI and there remain an appreciable number of patients at risk for restenosis. Use of systemic pharmacological therapy to inhibit coronary stent restenosis of bare metal stent has been largely unsuccessful. We have reported that erythropoietin could enhance reendothelialization leading to inhibition of in-stent restenosis by directly protecting endothelial apoptosis and mobilizing endothelial progenitors. The EPOC-AMI study is designed to assess the safety and the efficacy of systemic administration of erythropoietin aiming inhibition of neointimal hyperplasia after stent implantation in the patients with acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute myocardial infarction within 12hrs of symptom onset.
* Succeeded reperfusion due to primary PCI accomplished bare metal stent

Exclusion Criteria:

* Patients with cardiogenic shock (e.g. systolic BP<80mmHg,use of catecholamine, use of IABP)
* Patients with anemia required transfusion
* Patients who are unwilling or unable to comply with the trial protocol

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72

PRIMARY OUTCOMES:
In-stent Neointimal volume
In-stent Late lumen loss
Semi-Quantitative evaluation of infarcted size of myocardium

SECONDARY OUTCOMES:
left ventricular end diastolic volume
left ventricular end systolic volume
left ventricular ejection fraction
left ventricular wall motion index
binary restenosis
major adverse cardiac events (death,myocardial infarction, target lesion revascularization)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Matsubara, M.D., Ph.D., Study Chair — Kyoto Prefectural University of Medicine
Locations (1):
- Kyoto Prefectural University of Medicine, Kyoto, Kyoto, Japan

REFERENCES:
- [Background] Urao N, Okigaki M, Yamada H, Aadachi Y, Matsuno K, Matsui A, Matsunaga S, Tateishi K, Nomura T, Takahashi T, Tatsumi T, Matsubara H. Erythropoietin-mobilized endothelial progenitors enhance reendothelialization via Akt-endothelial nitric oxide synthase activation and prevent neointimal hyperplasia. Circ Res. 2006 Jun 9;98(11):1405-13. doi: 10.1161/01.RES.0000224117.59417.f3. Epub 2006 Apr 27. PMID 16645141
- [Derived] Taniguchi N, Nakamura T, Sawada T, Matsubara K, Furukawa K, Hadase M, Nakahara Y, Nakamura T, Matsubara H. Erythropoietin prevention trial of coronary restenosis and cardiac remodeling after ST-elevated acute myocardial infarction (EPOC-AMI): a pilot, randomized, placebo-controlled study. Circ J. 2010 Nov;74(11):2365-71. doi: 10.1253/circj.cj-10-0267. Epub 2010 Sep 8. PMID 20834185